CLINICAL TRIAL: NCT06574984
Title: Descriptive Study for Turoctocog Alfa Treatment Regimen in Iraqi Haemophilia A Patients - An Observational Retrospective Study
Brief Title: Study for Turoctocog Alfa Treatment Regimen in Iraqi Haemophilia A Patients
Status: Recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7008-7871
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Turoctocog alfa: Participants received turoctocog alfa intravenously.
  Interventions: Drug: Turoctocog alfa

INTERVENTIONS:
Drug: Turoctocog alfa — Turoctocog alfa was administered intravenously.
  Other Names: NovoEight

SUMMARY:
The study has descriptive purposes, with aim of assessing how turoctocog alfa is used in the everyday practice and to provide a baseline for the management of haemophilia A and does not involve any change in the clinical management of participants. Data will be extrapolated from the existing paper based medical records and uploaded to an electronic database specifically created for the study. Baseline information/history will be recorded at time of switching from previous FVIII replacement therapy to turoctocog alfa from the enrolled participants and outcomes will be collected according to participants visit format.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric and adult male patients
* On-demand and prophylactic patients with haemophilia A (any severity)
* Only previously treated patients (previous FVIII replacement therapy) will be included in the study

Exclusion Criteria:

* Patients diagnosed with coagulation disorders other than haemophilia A such as Von Willebrand disease
* Patients with documented presence of any FVIII inhibitor

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Participants received Turoctocog alfa intravenously.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Annual bleeding Rate (ABRs) among patients treated with different regimen of turoctocog alfa after previous FVIII replacement therapy | From baseline (first day of receiving turoctocog alpha) to month 12 after switching to turoctocog alfa
  Measured as count of all reported bleeding events divided by the number of months in the reporting time window (8 weeks to 12 months) and multiplied by 12.

SECONDARY OUTCOMES:
ABRs among patients treated with different regimen of turoctocog alfa after previous FVIII replacement therapy | From baseline (first day of receiving turoctocog alpha) to month 12 after switching to turoctocog alfa
  Measured as number of all reported bleeding events divided by the number of months in the reporting time window (8 weeks to 12 months) and multiplied by 12 across 4 age segments ( less than [<] 8 years, 8-14 years, 15-18 years, greater than [>] 18 years).
Change of primary prophylaxis regimen | From baseline (first day of receiving turoctocog alpha) to month 12 after switching to turoctocog alfa
  Measured as Yes/No.
Dose of turoctocog alfa | At month 12 after switching to turoctocog alfa
  Measured as international uniit per kilogram (IU/kg).
Haemostatic response to turoctocog alfa | At baseline and at month 12
  Measured as excellent, good, moderate, none.
Spontaneous ABR | At month 12 after switching to turoctocog alfa
  Measured as number of reported spontaneous bleeding events divided by the number of months in the reporting time window (8 weeks to 12 months) and multiplied by 12.
Annualized joint bleed rate (AJBR) | At month 12 after switching to turoctocog alfa
  Measured as number of reported joint bleeding episodes divided by the observation period in months multiplied by 12.
New target joint | At month 12 after switching to turoctocog alfa
  Measured as number resolution (Yes/No) affected joints.
Severity of bleeding | At month 12 after switching to turoctocog alfa
  Measured as mild / moderate / severe.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (5):
- Iraq (5):
  - National centre for Hamophilia, Baghdad
  - Novo Nordisk Investigational Site, Baghdad
  - Basrah Haemoplhilia centre, Basra
  - Hilla Haemophilia centre, Hillah
  - Karbala Haemophilia centre, Karbala

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com